CLINICAL TRIAL: NCT05306808
Title: Feasibility and Efficacy Study of Multidisciplinary Breast Cancer Rehabilitation During Chemotherapy
Brief Title: Multidisciplinary Rehabilitation Programme for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/00140
Record Dates: First submitted 2021-06-07; First posted 2022-04-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will attend a program combing 24 sessions of physiotherapy and 10 sessions of educational class over 12 weeks. Participants in the control group will be asked to exercise on their own.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- center-based exercise (Experimental): Participants in intervention group will attend a program combining 24 sessions of physiotherapy and 10 sessions of educational class over 12 weeks.
  Interventions: Other: physiotherapy class
- exercise on his/her own (No Intervention): Participants in control group will be asked to exercise on their own, they will only attend 10 sessions of educational class over 12 weeks.

INTERVENTIONS:
Other: physiotherapy class — The supervised 1-hour group exercise class will be conducted twice a week, with a maximum of 8 patients in each class. Subjects will be given a home log for exercise recording. If subjects are unable to attend exercise class for any reason (eg., low counts or feeling unwell, etc.), they will be advised to continue xercises at home. On the day of one of the exercise classes each week, there will be an additional 1-hour group education/ discussion session which may be conducted by PT, OT, APN, dietician or medical social worker. Topics covered will include physical activity, management of fatigue, lymphoedema, neuropathy, brain fog, return to work, stress, nutrition, sexuality, psychosocial and caregiver issues. There will be 10 sessions of educational class in total for each subject.
  Arms: center-based exercise

SUMMARY:
The study recruits breast cancer survivors who are already on chemotherapy or are going to start chemotherapy. Subjects will be asked for their preference to attend physiotherapy and educational class (for intervention group) or decline for it (for control group).

For intervention group, subject will attend 24 sessions of physiotherapy (exercise class) and 10 sessions of educational class over 12 weeks. The supervised 1-hour group exercise class will be conducted twice a week. Educational class will be once a week, with topics covering physical activity, management of fatigue, lymphoedema, neuropathy, brain fog, return to work, stress, nutrition, sexuality, psychosocial and caregiver issues.

Subjects in control group will be asked to exercise on their own in the 12 weeks.

12 weeks later, all subjects will attend a 2-hour survivorship transitional class, with topics covering cancer surveillance and follow up, addressing fear of recurrence: symptom and support, neuropathy/ fatigue/physical impairment/ brain fog, physical activity and diet, screening for colorectal and cervical cancers, return to work and community resources. During the class, a screening questionnaire will be administered to identify further physical, rehabilitation and psychosocial needs and to triage these patients to relevant hospital and community services.

Outcome assessment will be done at pre-intervention, after intervention, 6 months and 1 year after the intervention.

DETAILED DESCRIPTION:
This study will be a mixed study of both quantitative and qualitative research to investigate the effect of the holistic program of combining patient education and intra chemotherapy on cancer survivorship.

80 breast cancer survivors will be recruited from National University Cancer Institute, Singapore (NCIS). Breast cancer survivors who are already on chemotherapy or are going to start chemotherapy will be recruited.

Subjects will be asked their preference to attend physiotherapy and educational class (for intervention group) or decline for it (for control group). The study is not randomized as challenges in subject recruitment are expected otherwise. Patients in intervention group will attend a program combining 24 sessions of physiotherapy and 10 sessions of educational class over 12 weeks. Subjects in control group will be asked to exercise on their own.

The first visit for both groups will be an individual evaluation session by physiotherapist (PT), occupational therapist (OT), and study coordinator. Baseline assessments of outcome measures will be performed during the visit. PT and OT will also prescribe an individualized home exercise program for subjects in both groups.

Subsequent visits for intervention group will be 24 sessions of physiotherapy (exercise class) and 10 sessions of educational class over 12 weeks. The supervised 1-hour group exercise class will be conducted twice a week, with a maximum of 8 patients in each class. Subjects will be given a home log for exercise recording. If subjects are unable to attend exercise class for any reason (eg., low counts or feeling unwell, etc.), they will be advised to continue exercises at home. On the day of one of the exercise classes each week, there will be an additional 1-hour group education/ discussion session which may be conducted by PT, OT, APN, dietician or medical social worker. Topics covered will include physical activity, management of fatigue, lymphoedema, neuropathy, brain fog, return to work, stress, nutrition, sexuality, psychosocial and caregiver issues. There will be 10 sessions of educational class in total for each subject.

After completing all exercise classes and educational classes for subjects in intervention group, or after12 weeks' home exercise for subjects in control group, all subjects in both group will attend a 2-hour survivorship transitional class, which will be held in groups of up to 10 subjects. During the class, the trainer (usually APN) will educate and provide an overview of breast cancer survivorship issues, seek to empower with self-assessment skills and provide cancer survivors with information on available community resources. The class seeks to reintegrate cancer survivors back to the community and will also serve as a platform to screen for and identify those with further psychosocial and rehabilitation needs and triage them accordingly to the relevant hospital or community resources. The topics that will be covered in education will include cancer surveillance and follow up, addressing fear of recurrence: symptom and support, neuropathy/ fatigue/physical impairment/ brain fog, physical activity and diet, screening for colorectal and cervical cancers, return to work and community resources. During the class, a screening questionnaire will be administered to identify further physical, rehabilitation and psychosocial needs and to triage these patients to relevant hospital and community services.

The subsequent 2 visits for both groups will be outcome assessment. One is after the survivorship transitional class, and the other one is at 1 year after the survivorship transitional class. Outcome measures will be administered by PT, OT, and study coordinator.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 21 - 80 years old;
2. Breast cancer patients before or already on the treatment of chemotherapy, targeted therapy, and/or radiotherapy;
3. Be able to provide consent and complete questionnaires;
4. Be able to walk independently in the community without use of gait aids.
5. Breast cancer patients who are suitable for exercise.

Exclusion Criteria:

1. Pregnant;
2. Uncontrolled hypertension (Resting BP >160/90 mm Hg), or history of recurring or persistent hypotension in the past 2 months;
3. History of recent myocardial infarction or unstable angina (within the past 6 months);
4. Significant valvular disease i.e. severe aortic stenosis and moderate-severe mitral regurgitation;
5. Patient with end stage organ disease (e.g. ESRF, end stage COPD);
6. Tumor infiltration of axial or weight-bearing bones with risk of pathological fractures or compression of the spinal cord;
7. Patient with recent stroke within the past 6 months;
8. With other neuromusculoskeletal disorders such as osteoarthritis of such severity as to limit ability to participate in group exercise classes;
9. Already participating in regular physical activity (150min of moderate or 75min of vigorous physical activity/week);
10. Deemed inappropriate by primary oncologists.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females will be recruited
Enrollment: 70 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | Week0
  distance covered in 6 minutes with comfortable walking speed
6 minute walk test | Week12
  distance covered in 6 minutes with comfortable walking speed
6 minute walk test | Month6
  distance covered in 6 minutes with comfortable walking speed
Frenchay Activities Index (FAI) | Week0
  measure of engagement in instrumental activities of daily living. The scale provides a summed score from 15-60. Higher FAI score indicates higher instrumental activities
Frenchay Activities Index (FAI) | Week12
  measure of engagement in instrumental activities of daily living. The scale provides a summed score from 15-60. Higher FAI score indicates higher instrumental activities
Frenchay Activities Index (FAI) | Month6
  measure of engagement in instrumental activities of daily living. The scale provides a summed score from 15-60. Higher FAI score indicates higher instrumental activities
Functional Assessment of Cancer Therapy scale (FACT)-fatigue | Week0
  Fatigue scale, All items are summed to create a single fatigue score with a range from 0 to 52. Higher score indicates better outcome.
Functional Assessment of Cancer Therapy scale (FACT)-fatigue | Week12
  Fatigue scale, All items are summed to create a single fatigue score with a range from 0 to 52. Higher score indicates better outcome.
Functional Assessment of Cancer Therapy scale (FACT)-fatigue | Month6
  Fatigue scale, All items are summed to create a single fatigue score with a range from 0 to 52. Higher score indicates better outcome.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Week0
  Measurement on quality of life. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Week12
  Measurement on quality of life. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Month6
  Measurement on quality of life. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Week0
  IPAQ assesses 3 types of physical activity undertaken across the 4 domains- leisure time physical activity; domestic and gardening (yard) activities; work-related physical activity; transport-related physical activity- in the previous 7 days. The 3 types of activity assessed are walking, moderate-intensity activities and vigorous-intensity activities. The result s is not reported in scales. Computation of the total score for the IPAQ-SF requires summation of the duration (in minutes) and frequency (days) of the 3 types of activities across the 4 domains. Higher result indicates higher physical activity in the last 7 days.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Week12
  IPAQ assesses 3 types of physical activity undertaken across the 4 domains- leisure time physical activity; domestic and gardening (yard) activities; work-related physical activity; transport-related physical activity- in the previous 7 days. The 3 types of activity assessed are walking, moderate-intensity activities and vigorous-intensity activities. The result s is not reported in scales. Computation of the total score for the IPAQ-SF requires summation of the duration (in minutes) and frequency (days) of the 3 types of activities across the 4 domains. Higher result indicates higher physical activity in the last 7 days.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Month6
  IPAQ assesses 3 types of physical activity undertaken across the 4 domains- leisure time physical activity; domestic and gardening (yard) activities; work-related physical activity; transport-related physical activity- in the previous 7 days. The 3 types of activity assessed are walking, moderate-intensity activities and vigorous-intensity activities. The result s is not reported in scales. Computation of the total score for the IPAQ-SF requires summation of the duration (in minutes) and frequency (days) of the 3 types of activities across the 4 domains. Higher result indicates higher physical activity in the last 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Effie Chew, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National Univerity Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Chandran G, Tang N, Ngo ELP, Huang S, Tong SI, Ong JX, Chew E. Comparing the efficacy of a multi-dimensional breast cancer rehabilitation programme versus a home-based exercise programme during adjuvant cancer treatment. BMC Cancer. 2024 Mar 21;24(1):361. doi: 10.1186/s12885-024-12080-5. PMID 38509471